CLINICAL TRIAL: NCT01691248
Title: DEFLECT-1: A Phase 3b Multi-Center, Double-Blind, Randomized, Placebo Controlled Study to Demonstrate the Safety and Efficacy of Fidaxomicin for Prophylaxis Against Clostridium Difficile-Associated Diarrhea in Adults Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Fidaxomicin Versus Placebo for Prophylaxis Against Clostridium Difficile-Associated Diarrhea in Adults Undergoing Hematopoietic Stem Cell Transplantation (MK-5119-001)
Acronym: DEFLECT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Optimer Pharmaceuticals LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 5119-001; OPT-80-302 (Other: Optimerpharma Study Number)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Clostridium Difficile-Associated Diarrhea (CDAD)
Keywords: Clostridium difficile; Clostridium difficile-Associated Diarrhea; Prophylaxis; Hematopoietic Stem Cell Transplantation
MeSH Terms: interventions — Fidaxomicin; OPT 80

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fidaxomicin (Active Comparator): 200 mg Fidaxomicin tablet once daily for no longer than 40 days
  Interventions: Drug: fidaxomicin
- Placebo (Placebo Comparator): Placebo tablet once daily for no longer than 40 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: fidaxomicin — Fidaxomicin 200 mg tablet once daily from the start (+/- 2 days) of condition (prior to transplantation) or at the time of Fluoroquinolone initiation. Study drug treatment will continue until 7 days after either neutrophil engraftment or the completion of any Fluoroquinolone antibiotic regimen (whichever occurs later).
  Study drug treatment will stop at onset of CDAD or no longer than 40 days of duration, even if other antibiotics are still administered or neutrophil engraftment extends beyond 40 days.
  Other Names: DIFICID; DIFICLIR; OPT-80; PAR-101
  Arms: Fidaxomicin
Drug: Placebo — Placebo tablet once daily from the start (+/- 2 days) of condition (prior to transplantation) or at the time of Fluoroquinolone initiation. Treatment will continue until 7 days after either neutrophil engraftment or the completion of any Fluoroquinolone antibiotic regimen (whichever occurs later).
  Treatment will stop at onset of CDAD or no longer than 40 days of duration, even if other antibiotics are still administered or neutrophil engraftment extends beyond 40 days.
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate the efficacy and safety of Fidaxomicin versus placebo for prophylaxis against Clostridium difficile-Associated Diarrhea (CDAD) in adult participants undergoing hematopoietic stem cell transplantation (HSCT). The primary hypothesis is that Fidaxomicin is superior to placebo in preventing CDAD in participants undergoing HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older.
* Females of childbearing potential must be using an adequate and reliable method of contraception (e.g., abstinence, barrier with additional spermicide foam or jelly, intrauterine device, hormonal contraception). Males and females must agree to avoid conception during treatment and for four weeks following the end of study treatment.
* Is undergoing HSCT with planned Fluoroquinolone prophylaxis.
* Informed consent is provided.

Exclusion Criteria:

* Ongoing active CDAD infection (as evidenced by clinical signs of diarrhea along with the presence of either toxin A and/or B [or their respective genes, tcdA and/or tcdB] of C. difficile in the stool) or current treatment for CDAD.
* Undergoing cord blood transplants.
* Has fulminant colitis, toxic megacolon, or ileus.
* A history of inflammatory bowel disease (ulcerative colitis or Crohn's disease).
* Women who are pregnant or are actively breast feeding (all women of childbearing potential must have a negative pregnancy test result prior to dosing study drug).
* Use of any drugs potentially useful in the treatment of CDAD (e.g. oral Vancomycin, Metronidazole, oral Bacitracin, Fusidic Acid, Rifaximin, and Nitazoxanide).
* Any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant in the study, would make it unlikely for the participant to complete the study, or would confound the results of the study.
* Participation in other clinical research studies utilizing an investigational agent within one month prior to screening and during the study treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2012-10-10 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2015-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] de Almeida C, Wong M, Kleijn HJ, Wrishko RE. Predicted Bezlotoxumab Exposure in Patients Who Have Received a Hematopoietic Stem Cell Transplant. Clin Ther. 2023 Apr;45(4):356-362. doi: 10.1016/j.clinthera.2023.02.006. Epub 2023 Mar 9. PMID 36906440
- [Derived] Mullane KM, Winston DJ, Nooka A, Morris MI, Stiff P, Dugan MJ, Holland H, Gregg K, Adachi JA, Pergam SA, Alexander BD, Dubberke ER, Broyde N, Gorbach SL, Sears PS. A Randomized, Placebo-controlled Trial of Fidaxomicin for Prophylaxis of Clostridium difficile-associated Diarrhea in Adults Undergoing Hematopoietic Stem Cell Transplantation. Clin Infect Dis. 2019 Jan 7;68(2):196-203. doi: 10.1093/cid/ciy484. PMID 29893798

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fidaxomicin | Placebo
Started | 305 (Randomized) | 306 (Randomized)
Treated | 301 (Received at least 1 dose of study drug) | 299 (Received at least 1 dose of study drug)
Safety Analysis Set | 300 (A participant randomized to Fidaxomicin, received placebo instead.) | 300 (A participant randomized to Fidaxomicin, received placebo instead.)
Completed | 194 | 192
Not Completed | 111 | 114
Not completed — Protocol Violation | 43 | 27
Not completed — Adverse Event | 24 | 22
Not completed — Withdrawal by Subject | 20 | 18
Not completed — Confirmed CDAD | 14 | 31
Not completed — Lost to Follow-up | 2 | 5
Not completed — Reason not provided | 4 | 4
Not completed — Not Treated | 4 | 7

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) consisting of all randomized participants undergoing hematopoietic stem cell transplantation (HSCT) who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fidaxomicin | Placebo | Total
Number analyzed (Participants) | 301 | 299 | 600
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (12.00) | 55.1 (13.23) | 55.1 (12.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 103 | 228
  Male | 176 | 196 | 372

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Occurrence of CDAD From Start of Study Treatment up to 30 Days Post-treatment Follow-up.
Description: CDAD is defined as follows: Diarrhea: (change in bowel habits with >3 unformed bowel movements in a 24 hour period) and the presence of either toxin A and/or B (or their respective genes, tcdA and/or tcdB) of C. difficile in the stool determined by C. difficile toxin assay. Wald 95% Confidence Intervals (CI) are presented.
Time Frame: Up to 30 days post-treatment
Population: mITT consisting of all randomized participants undergoing HSCT who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fidaxomicin | Placebo
Number analyzed (Participants) | 301 | 299
Percentage of participants | 28.6 [23.5 to 33.7] | 30.8 [25.5 to 36.0]
Statistical Analysis 1: Comparison: Fidaxomicin vs Placebo; Test type: Superiority or Other; p = 0.2778, One-sided Wald p-value — 1-sided Wald test for a difference in proportions using an unpooled estimate of variance; Percentage Difference = 2.2, 95% CI 2-sided [-5.1 to 9.5] — Placebo minus Fidaxomicin

2. Secondary Outcome: Percentage of Participants With Occurrence of CDAD From Start of Study Treatment up to 60 Days Post-treatment.
Description: as for outcome 1
Time Frame: Up to 60 days post-treatment
Population: mITT consisting of all randomized participants undergoing HSCT who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fidaxomicin | Placebo
Number analyzed (Participants) | 301 | 299
Percentage of participants | 35.2 [29.8 to 40.6] | 35.8 [30.4 to 41.2]
Statistical Analysis 1: Comparison: Fidaxomicin vs Placebo; Test type: Superiority or Other; p = 0.4420, One-sided Wald p-value — 1-sided Wald test for a difference in proportions using an unpooled estimate of variance; Percentage difference = 0.6, 95% CI 2-sided [-7.1 to 8.2] — Placebo minus Fidaxomicin

3. Secondary Outcome: Percentage of Participants With Occurrence of CDAD From Start of Study Treatment up to Day 70 of Study.
Description: as for outcome 1
Time Frame: Up to Day 70 of study
Population: mITT consisting of all randomized participants undergoing HSCT who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Fidaxomicin | Placebo
Number analyzed (Participants) | 301 | 299
Percentage of participants | 29.2 [24.1 to 34.4] | 31.1 [25.9 to 36.4]
Statistical Analysis 1: Comparison: Fidaxomicin vs Placebo; Test type: Superiority or Other; p = 0.3091, One-sided Wald p-value — 1-sided Wald test for a difference in proportions using an unpooled estimate of variance; Percentage difference = 1.9, 95% CI 2-sided [-5.5 to 9.2] — Placebo minus Fidaxomicin

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (AEs) up to 32 days post treatment. Serious AEs (SAEs) up to 62 days post treatment.
Description: Participants who received at least one dose of study drug. One participant randomized to Fidaxomicin, received placebo instead.
Arm/Group | Fidaxomicin | Placebo
Serious Adverse Events (participants affected / at risk) | 98/300 | 92/300
Other Adverse Events (participants affected / at risk) | 297/300 | 298/300
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=300) | Placebo (N=300)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 17 (18) | 14 (14)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 1 (3)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Blindness (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1)
Inflammation (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 3 (3)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 5 (5) | 10 (10)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal hypertension (Hepatobiliary disorders) | 1 (1) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Acute graft versus host disease (Immune system disorders) | 3 (3) | 1 (1)
Acute graft versus host disease in intestine (Immune system disorders) | 0 (0) | 2 (2)
Acute graft versus host disease in skin (Immune system disorders) | 0 (0) | 1 (1)
Engraftment syndrome (Immune system disorders) | 1 (1) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 1 (1)
Graft versus host disease in intestine (Immune system disorders) | 2 (2) | 3 (3)
Graft versus host disease in lung (Immune system disorders) | 0 (0) | 1 (1)
Graft versus host disease in skin (Immune system disorders) | 2 (2) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Aspergillosis (Infections and infestations) | 1 (1) | 0 (0)
BK virus infection (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 3 (3) | 2 (3)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis gangrenous (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 4 (4) | 2 (2)
Cytomegalovirus viraemia (Infections and infestations) | 2 (2) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 1 (1)
Human herpesvirus 6 infection (Infections and infestations) | 0 (0) | 2 (2)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 4 (4)
Septic shock (Infections and infestations) | 1 (1) | 5 (5)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 4 (4)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Viraemia (Infections and infestations) | 0 (0) | 1 (1)
Viral haemorrhagic cystitis (Infections and infestations) | 2 (2) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug dispensing error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transplant failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood albumin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fluid imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral T-cell lymphoma unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 2 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure acute (Renal and urinary disorders) | 8 (9) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Haemodynamic instability (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 0 (0)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fidaxomicin (N=300) | Placebo (N=300)
Anaemia (Blood and lymphatic system disorders) | 40 (63) | 36 (52)
Febrile neutropenia (Blood and lymphatic system disorders) | 128 (131) | 98 (107)
Neutropenia (Blood and lymphatic system disorders) | 31 (63) | 40 (65)
Thrombocytopenia (Blood and lymphatic system disorders) | 54 (77) | 46 (77)
Sinus tachycardia (Cardiac disorders) | 13 (14) | 16 (16)
Tachycardia (Cardiac disorders) | 30 (39) | 43 (59)
Abdominal distension (Gastrointestinal disorders) | 16 (17) | 12 (14)
Abdominal pain (Gastrointestinal disorders) | 62 (71) | 63 (83)
Abdominal pain upper (Gastrointestinal disorders) | 20 (20) | 16 (24)
Constipation (Gastrointestinal disorders) | 55 (59) | 88 (107)
Diarrhoea (Gastrointestinal disorders) | 211 (286) | 220 (340)
Dry mouth (Gastrointestinal disorders) | 22 (24) | 32 (34)
Dyspepsia (Gastrointestinal disorders) | 44 (47) | 33 (35)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 15 (15) | 18 (19)
Haemorrhoids (Gastrointestinal disorders) | 18 (18) | 26 (27)
Nausea (Gastrointestinal disorders) | 184 (252) | 201 (284)
Oesophagitis (Gastrointestinal disorders) | 29 (29) | 24 (25)
Stomatitis (Gastrointestinal disorders) | 68 (89) | 75 (103)
Vomiting (Gastrointestinal disorders) | 119 (174) | 123 (172)
Asthenia (General disorders) | 22 (31) | 38 (47)
Chills (General disorders) | 28 (33) | 31 (39)
Fatigue (General disorders) | 117 (138) | 118 (149)
Mucosal inflammation (General disorders) | 107 (128) | 106 (134)
Oedema peripheral (General disorders) | 78 (99) | 63 (74)
Pyrexia (General disorders) | 69 (83) | 91 (103)
Oral candidiasis (Infections and infestations) | 17 (17) | 15 (15)
Aspartate aminotransferase increased (Investigations) | 12 (15) | 17 (24)
Blood creatinine increased (Investigations) | 13 (16) | 21 (23)
Haemoglobin decreased (Investigations) | 7 (11) | 16 (33)
Platelet count decreased (Investigations) | 17 (26) | 21 (31)
Decreased appetite (Metabolism and nutrition disorders) | 97 (117) | 106 (127)
Fluid overload (Metabolism and nutrition disorders) | 30 (30) | 29 (31)
Hyperglycaemia (Metabolism and nutrition disorders) | 13 (17) | 21 (27)
Hypocalcaemia (Metabolism and nutrition disorders) | 21 (25) | 13 (18)
Hypokalaemia (Metabolism and nutrition disorders) | 45 (53) | 44 (52)
Hypomagnesaemia (Metabolism and nutrition disorders) | 51 (68) | 51 (55)
Hypophosphataemia (Metabolism and nutrition disorders) | 37 (39) | 27 (28)
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 (21) | 25 (29)
Back pain (Musculoskeletal and connective tissue disorders) | 33 (37) | 40 (46)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (10) | 16 (20)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 (34) | 29 (31)
Dizziness (Nervous system disorders) | 44 (53) | 40 (43)
Dysgeusia (Nervous system disorders) | 31 (37) | 33 (36)
Headache (Nervous system disorders) | 75 (91) | 87 (105)
Neuropathy peripheral (Nervous system disorders) | 22 (24) | 7 (7)
Tremor (Nervous system disorders) | 17 (17) | 10 (11)
Anxiety (Psychiatric disorders) | 47 (54) | 39 (42)
Confusional state (Psychiatric disorders) | 16 (16) | 9 (10)
Insomnia (Psychiatric disorders) | 58 (61) | 62 (67)
Dysuria (Renal and urinary disorders) | 21 (22) | 23 (25)
Haematuria (Renal and urinary disorders) | 12 (13) | 16 (16)
Renal failure acute (Renal and urinary disorders) | 22 (22) | 23 (30)
Cough (Respiratory, thoracic and mediastinal disorders) | 43 (48) | 54 (60)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 (45) | 30 (34)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 20 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 24 (29)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 19 (19)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 18 (18)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 43 (47) | 42 (49)
Alopecia (Skin and subcutaneous tissue disorders) | 17 (19) | 12 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 20 (21) | 23 (26)
Erythema (Skin and subcutaneous tissue disorders) | 18 (19) | 10 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 32 (38) | 32 (36)
Rash (Skin and subcutaneous tissue disorders) | 52 (63) | 46 (55)
Rash generalised (Skin and subcutaneous tissue disorders) | 7 (8) | 18 (20)
Hypertension (Vascular disorders) | 35 (38) | 40 (50)
Hypotension (Vascular disorders) | 43 (53) | 48 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication or other public presentation of results from this study requires prior review and written approval of the Sponsor. Draft abstracts, manuscripts, and materials for presentation at scientific meetings should be provided to the Sponsor at least 90 working days prior to abstract or other relevant submission deadlines.